CLINICAL TRIAL: NCT04236700
Title: Oral and Buccal Evaluation of Mobile Beach Workers
Brief Title: Buccal Evaluation of Mobile Beach Workers
Status: Recruiting | Type: Observational
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS G. ROMAN TORRES, Professor, Universidade Metropolitana de Santos
Other Study IDs: SantosMU7
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Buccal Cavity Cancer; Labial Lipoma
Keywords: Buccal cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- beach workers: Workers must undergo clinical examinations of the upper and lower lips, performed by previously calibrated researchers, through semi-technical inspection and palpation maneuvers, in order to identify injuries. Photo cameras can be used to improve the visibility of the lips using the image enhancement feature, to confirm the diagnosis. The clinical examination will include: dryness, atrophy, scaly lesions, lip swelling, erythema, ulcerations, cloudy demarcations between the vermilion of the lip and skin, demarcated folds along the lip, white spots or plaques, crusts, stained or pale areas.
  They should be evaluated with the application of a previously validated questionnaire containing information related to personal data, information on occupation and health was completed according to the responses of the volunteers. The OHIP-14 quality of life questionnaire will be applied together
  Interventions: Other: Oral clinical exam

INTERVENTIONS:
Other: Oral clinical exam — Detailed anamnesis, with information regarding the time of sun exposure, protection measures, medical history and application of questionnaires will be carried out. Dental dental and tissue examination should be performed

SUMMARY:
Tumors in the oral region occur more frequently in men over 40, but can affect people of both gender and all ages, even children. The prevention of oral cancer acquires relevance in public health, particularly if the investigators consider that the preventive approach is compatible with the nature of this disease, as the mouth favors easy visual access. The objective of this study is evaluation the prevalence of oral and perioral injuries in workers who were exposed to the sun on the beaches, investigating possible associations of a sociodemographic, occupational and general health nature.

DETAILED DESCRIPTION:
Tumors in the oral region occur more frequently in men over 40, but can affect people of both sexes and all ages, even children. The prevention of oral cancer acquires relevance in public health, particularly if the investigators consider that the preventive approach is compatible with the nature of this disease, as the mouth favors easy visual access. The objective of this study is evaluation the prevalence of oral and perioral injuries in workers who were exposed to the sun on the beaches, investigating possible associations of a sociodemographic, occupational and general health nature. Firstly, information about the care, symptoms and forms of prevention will be explained for each worker approached, if the individual agrees to an oral examination, it can be performed by evaluating lips and peri-oral mucosa and within the needs of oral treatment, it can be referred for treatment at the clinic of the Dentistry Especialist Center of Santos/SP The street vendors who underwent the first assessment will be visited 2 more times according to the schedule, after the carnival of 2020 being the last assessment and thus being able to have data on the effectiveness of the information and past care during the visits made. As expected results, a greater awareness of the dangers of sun exposure, greater protection care and the ability to carry out self-examination at home being an information disseminator.

ELIGIBILITY:
Inclusion Criteria:

* be walking beach worker

Exclusion Criteria:

* not wanting to participate in the evaluation

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample will consist of adult individuals of both sexes exposed to the sun directly and indirectly. The independent variables analyzed were: sex, age, income (in reais), years of study, type of work, frequency of weekly sun exposure, time of daily sun exposure, cumulative time of sun exposure and photoprotection measures at the occupational level. Health data will be collected on habits (alcoholism and smoking) and skin type, according to the Fitzpatrick classification
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
number of workers with labial injuries | 2 months
  beach workers who do not adopt protective measures may have tissue damage to their lips

CONTACTS AND LOCATIONS:
Overall Officials: CAIO VINICIUS G ROMAN TORRES, Principal Investigator — University of Santo Amaro
Locations (2):
- Brazil (2):
  - Caio Vinicius Gonçalves Roman Torres, Santos, São Paulo
  - Caio Torres, Santos, São Paulo

IPD SHARING:
Plan to Share IPD: No
The collected data will be imported into the Stata 10.0 software platform. Descriptive analysis of all data related to dependent and independent variables, chi-square statistical tests and calculation of prevalence ratios and the respective confidence intervals. The multiple analysis will be performed using the robust Poisson regression by the hybrid method parameter to estimate the prevalence rates of lip lesions adjusted for sex, age, type of work, photo-protection measures, use of lip protector, use of cap / hat, skin type, any habit (smoking or drinking). The significance level of 5% will be adopted for all tests.

REFERENCES:
- [Result] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Result] Campisi G, Margiotta V. Oral mucosal lesions and risk habits among men in an Italian study population. J Oral Pathol Med. 2001 Jan;30(1):22-8. doi: 10.1034/j.1600-0714.2001.300104.x. PMID 11140896
- [Result] English DR, Armstrong BK, Kricker A, Fleming C. Sunlight and cancer. Cancer Causes Control. 1997 May;8(3):271-83. doi: 10.1023/a:1018440801577. PMID 9498892